CLINICAL TRIAL: NCT03297502
Title: Multicenter Study of the Safety and Bioequivalence of Par's Pimecrolimus Cream, 1% and RLD Elidel® (Pimecrolimus Cream, 1%) and Compare Both Active Treatments to a Vehicle Control in Treatment of Mild to Moderate Atopic Dermatitis
Brief Title: Safety and Bioequivalence of Pimecrolimus Cream 1% and Elidel R in Treatment of Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYM 2016-01
Record Dates: First submitted 2017-09-22; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pimecrolimus cream, 1% (Experimental)
  Interventions: Drug: pimecrolimus cream 1%
- Elidel (pimecrolimus) cream 1% (Active Comparator)
  Interventions: Drug: Elidel (pimecrolimus) cream 1%
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pimecrolimus cream 1%
  Arms: Pimecrolimus cream, 1%
Drug: Elidel (pimecrolimus) cream 1%
  Arms: Elidel (pimecrolimus) cream 1%
Drug: placebo
  Arms: placebo

SUMMARY:
A phase 3, double-blind, randomized, parallel-group, placebo-controlled, multicenter study to evaluate the safety and bioequivalence of Par Pharmaceutical Inc.'s Pimecrolimus Cream, 1% and Reference Listed Elidel® (Pimecrolimus Cream, 1%). The study compares both active treatments to a placebo control in the treatment of mild to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent/assent for the study.
2. Non-immunocompromised male or female aged 12 years or older.
3. A clinical diagnosis of mild to moderate atopic dermatitis that has failed to respond adequately to other topical prescription treatments for atopic dermatitis, or subjects for whom the use of those other treatments is deemed inadvisable.
4. A diagnosis of atopic dermatitis for at least 3 months.
5. A baseline Investigator's Global Assessment (IGA) of disease severity of mild or moderate (score of 2 or 3). (See Section 9.6.10 for the scale.)
6. An affected area of atopic dermatitis involvement of at least 5% of the body surface area (BSA) at Visit 2/Day 1 (Baseline), as defined by the criteria of Hanifin and Rajka (1980).
7. Treatment with a bland emollient for at least 7 days prior to Visit 2/Day 1 (Baseline).
8. Agree to adhere to protocol-specified requirements and concomitant therapy restrictions.
9. Willing to avoid constant sun exposure and the use of tanning booths or other UV light sources during participation in the study.
10. In general good health, non-immunocompromised, and free from any clinically significant disease, other than atopic dermatitis, that might interfere with the study evaluations.
11. Willing and able to understand and comply with the requirements of the study, apply the study medication as instructed, return for the required study visits, comply with therapy prohibitions, and complete the study.
12. Female subjects of childbearing potential (excluding women who are surgically sterilized [hysterectomy, bilateral tubal ligation, or bilateral ovariectomy] or have been postmenopausal for at least 1 year) must have a negative urine pregnancy test and must be willing to use a medically accepted method of contraception during the study. The following are considered acceptable methods of birth control for the purpose of this study: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device (IUD), hormonal IUD (Mirena®), Essure® permanent birth control, and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active.

Exclusion Criteria:

1. Females who are pregnant, breastfeeding, intending to become pregnant during the study, or who do not agree to use an acceptable form of birth control during the study.
2. Active cutaneous bacterial or viral infection in any proposed treatment area at Visit 2/Baseline (e.g., clinically infected atopic dermatitis).
3. Sunburn, extensive scarring, or pigmented lesion(s) in any treatment area at Visit 2/Baseline that would interfere with the study evaluations.
4. History of confounding skin conditions, e.g., psoriasis, rosacea, erythroderma, or ichthyosis.
5. History or presence of Netherton's Syndrome, immunological deficiencies or diseases, HIV, diabetes, malignancy, serious active or recurrent infection, clinically significant severe renal insufficiency, or severe hepatic disorders.
6. Use of any treatment listed in Table 9.1 more recently than the indicated washout period prior to Visit 2/Baseline.
7. Need or intent to continue to use any treatment listed in Table 9.1 during the current study.

   Table 9.1 Medications, Supplements, and Other Substances Prohibited for Study Entry Prohibited Medications, Supplements, and Other Substances Washout Period Prior to Randomization Visit 2/Baseline
   * Systemic corticosteroids (oral and injectable [intravenous and intramuscular]) (Intranasal and Inhalational steroids are allowed if use is kept constant during the study)
   * UVA/UVB therapy
   * PUVA (psoralen plus ultraviolet A) therapy
   * Tanning booths
   * Nonprescription UV light sources
   * Immunomodulators or immunosuppressive therapies
   * Interferon
   * Cytotoxic drugs (e.g., methotrexate, cyclophosphamide, azathioprine)
   * Oral retinoids
   * Systemic anti-fungals
   * Tacrolimus
   * Pimecrolimus 30 days (1 month)
   * Systemic antibiotics
   * Topical calcipotriene or other topical vitamin D preparations
   * Topical retinoids 14 days (2 weeks)
   * Topical and oral antihistamines
   * Topical antibiotics
   * Topical corticosteroids
   * Topical antifungals
   * Other topical drug products 7 days (1 week)
   * Any topical product (e.g., sunscreens, lotions, creams) in areas to be treated except for bland emollient (moisturizer)
   * Grapefruit or grapefruit juice which is considered a CYP3A inhibitor 24 hours
8. Current use of calcium channel blockers (e.g, amlodipine, nifedipine, verapamil, diltiazem, felodipine, isradipine, nisoldipine, etc) and/or cimetidine (e.g., Tagamet) which are CPY3A inhibitors.
9. Known allergy or hypersensitivity to pimecrolimus or any other component of the Test or Reference product.
10. Unwilling to minimize or avoid natural and artificial sunlight exposure during treatment.
11. Consumption of excessive alcohol, abuse of drugs, or a condition that could compromise the subject's ability to comply with study requirements.
12. Any clinically significant condition or situation other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.
13. Use of any investigational drug or investigational device within 30 days prior to Visit 2/Baseline.
14. Previous participation in this study.
15. Employees of the research center or investigator.
16. Family members of employees of the research center or investigator.
17. Family members living in the same household participating at the same time.

Table 9.2 Medications (Prescription and Over-the-Counter), Supplements, and Other Substances Prohibited During the Study Prohibited Medications, Supplements, and Other Substances Treatment for atopic dermatitis other than assigned study medication or bland emollient.

Topical or systemic (oral and injectable) corticosteroid (Intranasal and inhalational steroids are allowed if kept constant during the study) Topical or systemic antibiotic Topical or systemic antifungal Topical or oral antihistamine (e.g., diphenhydramine, hydroxyzine) Immunosuppressive drugs Immunomodulator (e.g., tacrolimus) Calcipotriene or other topical vitamin D preparations Topical or oral retinoids Interferon Cyclosporine Methotrexate Azathioprine CPY3A inhibitor (e.g., erythromycin, itraconazole, ketoconazole, fluconazole, calcium channel blockers, cimetidine, grapefruit or grapefruit juice) Topical product other than assigned study medication or bland emollient (e.g., sunscreen, new brand of cosmetic or cleanser, cream, lotion, ointment, or powder) applied on or near the treatment area(s) Phototherapy (e.g., PUVA, UVA or UVB therapy)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with treatment success in each treatment group | Day 15
  Treatment success is defined as an Investigator's Global Assessment (IGA) Rating of "clear" or "almost clear" ( i.e., a score of 0 or 1 on a scale of 0 [clear] through 4. IGA Scale: 0 = Clear (minor discoloration, no erythema, induration, population, oozing/crusting. 1= Almost Clear (trace, faint erythema, almost no induration/population, no oozing/crusting. 2 = Mild (faint erythema, mild induration/population, no oozing/crusting. 3 = Moderate (Pink-red erythema, moderate induration/population, some oozing/crusting. 4 = Severe (Deep/bright erythema, severe induration/population, with oozing/crusting.

SECONDARY OUTCOMES:
Change from baseline in severity (erythema) | Baseline, Day 15
  Change from baseline in severity in clinical signs and symptoms of erythema is assessed.
  0 = None: No erythema present
  1. = Mild: Slight erythema, very light-pink
  2. = Moderate: Dull red, clearly distinguishable
  3. = Severe: Deep/dark red
Change from baseline in severity (induration/population) | Baseline, Day 15
  Change from baseline in severity in clinical signs and symptoms of induration/papulation is assessed.
  0 = None: No elevation
  1. = Mild: Slightly perceptible elevation
  2. = Moderate: Clearly perceptible elevation
  3. = Severe: Marked and extensive elevation
Change from baseline in severity (lichenification) | Baseline, Day 15
  Change from baseline in severity in clinical signs and symptoms of lichenification is assessed.
  0 = None: No lichenification
  1. = Mild: Slight thickening of the skin discernible only by touch and with skin markings minimally exaggerated
  2. = Moderate: Definite thickening of the skin with skin markings exaggerated so that they form a visible criss-cross pattern
  3. = Severe: Thickened indurated skin with skin markings visibly portraying an exaggerated criss-cross pattern
Change from baseline in severity (pruritis) | Baseline, Day 15
  Change from baseline in severity in clinical signs and symptoms of puritus is assessed.
  0 = None: No itching
  1. = Mild: Occasional, slight itching/scratching
  2. = Moderate: Constant or intermittent itching/scratching/discomfort that is not disturbing sleep
  3. = Severe: Bothersome itching/scratching/discomfort that is disturbing sleep

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, RPh, Study Director — Endo Pharmaceuticals